CLINICAL TRIAL: NCT04821063
Title: A Randomized, Partially Double-Blind, Four-Period, Four-Treatment, Crossover Study Investigating the Placebo-Corrected Effects of a Therapeutic Dose (100 mg) and a Supratherapeutic Dose (300 mg) of ITF2357 (Givinostat) and Moxifloxacin on QT/QTC Interval in Healthy Male and Female Subjects
Brief Title: Placebo-Corrected Effects of Therapeutic Dose (100 mg) and Supratherapeutic Dose (300 mg) of ITF2357 (Givinostat) and Moxifloxacin on QT/QTC Interval
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Italfarmaco (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ITF/2357/54; 2020-003105-63 (EudraCT Number)
Record Dates: First submitted 2021-03-26; First posted 2021-03-29 (Actual); Results first posted 2024-01-11 (Actual); Last update posted 2024-01-11 (Actual); Status verified 2023-04

CONDITIONS: Duchenne and Becker Muscular Dystrophy; Polycytemia Vera
MeSH Terms: conditions — Muscular Dystrophy, Duchenne | interventions — givinostat hydrochloride; givinostat; Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: ITF2357 (therapeutic dose and supratherapeutic dose, and placebo) will be administered in a double-blinded fashion whereas no blinding will be needed with treatment moxifloxacin.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Therapeutic dose: ITF2357 100 mg (Experimental): Participants will receive a single dose of ITF2357 100 mg administered as 10 milliliters (mL) of ITF2357 10 milligrams per milliliter (mg/mL) oral suspension and 20 mL of placebo matched to ITF2357 oral suspension under fasting conditions on Day 1 of respective period as per the assigned treatment sequence.
  Interventions: Drug: ITF2357 10 mg/mL; Drug: Placebo
- Supratherapeutic dose: ITF2357 300 mg (Experimental): Participants will receive a single dose of ITF2357 300 mg administered as 30 mL of ITF2357 10 mg/mL oral suspension under fasting conditions on Day 1 of respective period as per the assigned treatment sequence.
  Interventions: Drug: ITF2357 10 mg/mL
- Placebo (Placebo Comparator): Participants will receive a single dose of placebo matched to ITF2357 administered as 30 mL oral suspension under fasting conditions on Day 1 of respective period as per the assigned treatment sequence.
  Interventions: Drug: Placebo
- Moxifloxacin (Active Comparator): Participants will receive a single dose of moxifloxacin 400 mg tablet under fasting conditions on Day 1 of respective period as per the assigned treatment sequence.
  Interventions: Drug: Moxifloxacin Hydrochloride

INTERVENTIONS:
Drug: ITF2357 10 mg/mL — Dose: 100 mg (administered as 10 mL); Dosage form: suspension; Route of administration: oral
  Other Names: Givinostat
  Arms: Therapeutic dose: ITF2357 100 mg
Drug: ITF2357 10 mg/mL — Dose: 300 mg (administered as 30 mL); Dosage form: suspension; Route of administration: oral
  Other Names: Givinostat
  Arms: Supratherapeutic dose: ITF2357 300 mg
Drug: Placebo — Dose: 20 mL; Dosage form: suspension; Route of administration: oral
  Arms: Therapeutic dose: ITF2357 100 mg
Drug: Moxifloxacin Hydrochloride — Dose: 400 mg; Dosage form: tablet; Route of administration: oral
  Arms: Moxifloxacin
Drug: Placebo — Dose: 30 mL; Dosage form: suspension; Route of administration: oral
  Arms: Placebo

SUMMARY:
The study will evaluate the effect of a therapeutic dose and a supratherapeutic dose of ITF2357 on the QT/QTc interval.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, non-smoker (no use of tobacco or nicotine products within 3 months prior to screening), greater than or equal to (>=) 18 and less than or equal to (<=) 55 years of age, with body mass index (BMI) greater than (>) 18.5 and less than (<) 30.0 kilograms per meter square (kg/m^2) and body weight >=55 kilograms (kg) and <=100 kg for females and body weight >=60 kg and <=100 kg for males.
2. Healthy as defined by:

   1. The absence of clinically significant illness and major surgery within 4 weeks prior to dosing. Participants vomiting within 24 hours pre-dose will be carefully evaluated for upcoming illness/disease. Inclusion pre-dosing of the patient in the study is at the discretion of the Investigator, depending on his/her clinical judgement.
   2. The absence of clinically significant history of neurological, endocrinal, cardiovascular, pulmonary, hematological, immunologic, psychiatric, gastrointestinal, renal, hepatic, and metabolic disease.
3. Non-childbearing potential female defined as:

   1. Post-menopausal female (absence of menses for 12 months prior to the first study drug administration, bilateral oophorectomy or hysterectomy with bilateral oophorectomy at least 6 months prior to the first study drug administration); or
   2. Surgically sterile female (hysterectomy or tubal ligation at least 6 months prior to drug administration).
4. Females of childbearing potential who are sexually active with a male partner must be willing to use one of the following acceptable contraceptive methods throughout the study and for at least 90 days after the last study drug administration:

   1. Simultaneous use of intra-uterine contraceptive device, without hormone release system placed at least 4 weeks prior to study drug administration, and condom for the male partner;
   2. Simultaneous use of diaphragm or cervical cap with intravaginally applied spermicide and male condom for the male partner, started at least 21 days prior to study drug administration;
5. Male participants who are not vasectomized for at least 6 months, and who are sexually active with a female partner of childbearing potential (childbearing potential females are defined as women that are neither post-menopausal nor surgically sterile) must be willing to use one of the following acceptable contraceptive methods from the first study drug administration until at least 90 days after the last study drug administration:

   1. Simultaneous use of a male condom and, for the female partner, hormonal contraceptives used since at least 4 weeks or intra-uterine contraceptive device placed since at least 4 weeks;
   2. Simultaneous use of a male condom and, for the female partner, a diaphragm or cervical cap with intravaginally applied spermicide.
6. Male participants (including men who have had a vasectomy) with a pregnant partner must agree to use a condom from the first study drug administration until at least 90 days after the last study drug administration.
7. Male participants must be willing not to donate sperm until 90 days following the last study drug administration.
8. Female participants must be willing not to donate ovules until 90 days following the last study drug administration.
9. Participant's written informed consent obtained prior to any study-related procedure.
10. Willingness and capability to comply with the requirements of the study and ability to understand the study procedures and the risks involved.
11. Willing to take out dentures and mouth piercings for study procedures.

Exclusion Criteria:

1. Any clinically significant abnormality at physical examination, clinically significant abnormal laboratory test results or positive test for human immunodeficiency virus (HIV), hepatitis B, or hepatitis C found during medical screening.
2. Clinically significant vital sign abnormalities (systolic blood pressure lower than 90 or over 140 millimeter of mercury [mmHg], diastolic blood pressure lower than 60 or over 90 mmHg, or heart rate less than 40 or over 100 beats per minute [bpm]) at screening. For eligibility purposes, not the mean value, but the two single measurements will be considered.
3. Any of the following abnormalities on 12-lead ECG at screening. PR (PR interval) >210 millisecond (msec); QRS (QRS complex) >120 msec; QTcF >450 msec; any abnormality of cardiac rhythm other than sinus arrhythmia; abnormality of T-wave morphology that will impair the ability to measure the QT interval reliably. The averaged value of three ECGs 5 minutes apart from each other will be used; evaluations have to be used for the evaluation of the QTc interval requested by this exclusion criteria.
4. Participants with history of sustained and non-sustained cardiac arrhythmias (ECG demonstrated), participants with a family history of sudden cardiac death and participants with a history of additional risk factors for TdP, heart failure, hypokalemia, LQTS).
5. Any of the following abnormal laboratory test values at screening or at baseline (Day -1) of Period 1:

   1. Platelet count <125*10^9 per liter (/L)
   2. Absolute neutrophil count <1.2*10^9/L
6. Participants who have cardiovascular condition such as, but not limited to unstable ischemic heart disease, New York Heart Association (NYHA) Class III/IV left ventricular failure, acute ischemic heart disease in the last year prior to study screening, which may impact the safety of the participant or the evaluation of the result of the study according to the Investigator's judgment; cardiovascular conditions should be discarded based on the results obtained on the ECG, medical examination and routine lab test.
7. Positive urine drug screen, alcohol breath test or urine cotinine test at screening or at baseline (Day -1).
8. History of anaphylaxis reaction or clinically significant drug hypersensitivity reaction (e.g., angioedema, Stevens-Johnson syndrome, Acute Generalized Exanthematous Pustulosis, Drug-induced hypersensitivity syndrome, Drug-induced neutropenia).
9. History of allergic reactions to ITF2357, histone deacetylases (HDAC) inhibitors, or other related drugs, moxifloxacin, other quinolones, or to any excipient in the formulation.
10. Positive pregnancy test at screening or at baseline (Day -1).
11. Participants with a sorbitol intolerance or sorbitol malabsorption or have fructose intolerance.
12. Current or recent (within 3 months of study drug administration) clinically significant gastrointestinal disease that can interfere with drug absorption.
13. Gastrointestinal surgery that interferes with physiological absorption and motility (i.e., gastric bypass, duodenectomy) or gastric bands.
14. History of significant alcohol abuse within 1 year prior to screening or regular use of alcohol within 6 months prior to the screening visit (more than 14 units of alcohol per week [1 unit = 150 milliliter [mL] of wine, 360 mL of beer, or 45 mL of 40 percent [%] alcohol]).
15. History of significant drug abuse within 1 year prior to screening or use of soft drugs (such as marijuana) within 3 months prior to the screening visit or hard drugs (such as cocaine, phencyclidine [PCP], crack, opioid derivatives including heroin, and amphetamine derivatives) within 1 year prior to screening.
16. Use of ITF2357 for a medical condition or in the context of another clinical trial within a period of 30 days prior to the first dosing.
17. Participation in a clinical research study involving the administration of an investigational or marketed drug or device within 30 days prior to the first dosing, administration of a biological product in the context of a clinical research study within 90 days prior to the first dosing, or concomitant participation in an investigational study involving no drug or device administration.
18. Use of medications for the timeframes specified below, with the exception of medications exempted by the Investigator on a case-by-case basis because they are judged unlikely to affect the pharmacokinetic profile of the study drug or participant safety (e.g., topical drug products without significant systemic absorption):

    1. Prescription medications within 14 days prior to the first dosing;
    2. OTC products (with the exception of the occasional use of acetaminophen [up to 2 grams [g] daily]) and natural health products (including herbal remedies, homeopathic and traditional medicines, probiotics, food supplements such as vitamins, minerals, amino acids, essential fatty acids, and protein supplements used in sports) within 7 days prior to the first dosing;
    3. Depot injection or implant of any drug within 3 months prior to the first dosing;
    4. Any drugs known to induce or inhibit hepatic drug metabolism (including St. John's wort) within 30 days prior to the first dosing.
19. Donation of plasma within 7 days prior to dosing. Donation or loss of blood (excluding volume drawn at screening) of 50 mL to 499 mL of blood within 30 days, or more than 499 mL within 56 days prior to the first dosing.
20. Breast-feeding participant.
21. Inability to be venipunctured and/or tolerate catheter venous access;
22. Inability or difficulty to swallow tablets or suspension.
23. Any reason which, in the opinion of the Investigator, would prevent the participant from participating in the study.
24. History or presence of other diseases, metabolic dysfunctions, physical examination findings, or any clinically relevant abnormal laboratory value at screening suggesting an unknown disease and requiring further clinical investigation or which may impact the safety of the participant or the evaluation of the result of the study according to the Investigator's judgment.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2021-04-13 (Actual); Primary Completion 2021-06-18 (Actual); Study Completion 2021-06-18 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Québec, Québec, Canada

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at a single center in Canada. A total of 34 healthy non-smoker were screened in the study, of which 31 participants were enrolled and received the study treatment. Screen failures were mainly due to not meeting inclusion criteria.
Pre-assignment Details: Participants were administered the following treatments: Treatment T (Therapeutic dose of ITF2357 100 mg), Treatment ST (Supratherapeutic dose of ITF2357 300 mg), Treatment P (Placebo), and Treatment M (Moxifloxacin) in 4-periods and 12-sequences in this study.
Groups:
- Sequence TSTPM: Participants received a single dose of ITF2357 100 mg (Treatment T) oral suspension under fasted condition in Period 1, followed by a single dose of ITF2357 300 mg (as 10 mg/mL, Treatment ST) oral suspension under fasted conditions in Period 2, followed by a single dose of placebo matched to ITL2357 (Treatment P) oral suspension under fasted conditions in Period 3, followed by a single dose of moxifloxacin hydrochloride 400 mg tablets (Treatment M) under fasted conditions in Period 4, on Day 1 in the treatment period. Each period was separated by a washout period of 7 days.
- Sequence STMTP: Participants received a single dose of ITF2357 300 mg (as 10 mg/mL, Treatment ST) oral suspension under fasted conditions in Period 1, followed by a single dose of moxifloxacin hydrochloride 400 mg tablets (Treatment M) under fasted conditions in Period 2, followed by a single dose of ITF2357 100 mg (Treatment T) oral suspension under fasted condition in Period 3, followed by a single dose of placebo matched to ITL2357 (Treatment P) oral suspension under fasted conditions in Period 4 on Day 1 in the treatment period. Each period was separated by a washout period of 7 days.
- Sequence PTMST: Participants received a single dose of placebo matched to ITL2357 (Treatment P) oral suspension under fasted conditions in Period 1, followed by a single dose of ITF2357 100 mg (Treatment T) oral suspension under fasted condition in Period 2, followed by a single dose of moxifloxacin hydrochloride 400 mg tablets (Treatment M) under fasted conditions in Period 3, followed by a single dose of ITF2357 300 mg (as 10 mg/mL, Treatment ST) oral suspension under fasted conditions in Period 4 on Day 1 in the treatment period. Each period was separated by a washout period of 7 days.
- Sequence MPSTT: Participants received a single dose of moxifloxacin hydrochloride 400 mg tablets (Treatment M) under fasted conditions in Period 1, followed by a single dose of placebo matched to ITL2357 (Treatment P) oral suspension under fasted conditions in Period 2, followed by a single dose of ITF2357 300 mg (as 10 mg/mL, Treatment ST) oral suspension under fasted conditions in Period 3, followed by a single dose of ITF2357 100 mg (Treatment T) oral suspension under the fasted condition in Period 4 on Day 1 in the treatment period. Each period was separated by a washout period of 7 days.
- Sequence STPTM: Participants received a single dose of ITF2357 300 mg (as 10 mg/mL, Treatment ST) oral suspension under fasted conditions in Period 1, followed by a single dose of placebo matched to ITL2357 (Treatment P) oral suspension under fasted conditions in Period 2, followed by a single dose of ITF2357 100 mg (Treatment T) oral suspension under fasted condition in Period 3, followed by a single dose of moxifloxacin hydrochloride 400 mg tablets (Treatment M) under fasted conditions in Period 4, on Day 1 in the treatment period. Each period was separated by a washout period of 7 days.
- Sequence PMSTT: Participants received a single dose of placebo matched to ITL2357 (Treatment Placebo [P]) oral suspension under fasted conditions in Period 1, followed by a single dose of moxifloxacin hydrochloride 400 milligrams (mg) tablets (Treatment M) under fasted conditions in Period 2, followed by a single dose of ITF2357 300 mg (as 10 mg/mL, Treatment ST) oral suspension under fasted conditions in Period 3, followed by a single dose of ITF2357 100 mg (Treatment T) oral suspension under the fasted condition in Period 4 on Day 1 in the treatment period. Each period was separated by a washout period of 7 days.
- Sequence TSTMP: Participants received a single dose of ITF2357 100 mg (Treatment T) oral suspension under fasted condition in Period 1, followed by a single dose of ITF2357 300 mg (as 10 mg/mL, Treatment ST) oral suspension under fasted conditions in Period 2, followed by a single dose of moxifloxacin hydrochloride 400 mg tablets (Treatment M) under fasted conditions in Period 3, followed by a single dose of placebo matched to ITL2357 (Treatment P) oral suspension under fasted conditions in Period 4 on Day 1 in the treatment period. Each period was separated by a washout period of 7 days.
- Sequence MTPST: Participants received a single dose of moxifloxacin hydrochloride 400 mg tablets (Treatment M) under fasted conditions in Period 1, followed by a single dose of ITF2357 100 mg (Treatment T) oral suspension under fasted condition in Period 2, followed by a single dose of placebo matched to ITL2357 (Treatment P) oral suspension under fasted conditions in Period 3, followed by a single dose of ITF2357 300 mg (as 10 mg/mL, Treatment ST) oral suspension under fasted conditions in Period 4 on Day 1 in the treatment period. Each period was separated by a washout period of 7 days.
- Sequence PTSTM: Participants received a single dose of placebo matched to ITL2357 (Treatment P) oral suspension under fasted conditions in Period 1, followed by a single dose of ITF2357 100 mg (Treatment T) oral suspension under fasted condition in Period 2, followed by a single dose of ITF2357 300 mg (as 10 mg/mL, Treatment ST) oral suspension under fasted conditions in Period 3, followed by a single dose of moxifloxacin hydrochloride 400 mg tablets (Treatment M) under fasted conditions in Period 4, on Day 1 in the treatment period. Each period was separated by a washout period of 7 days.
- Sequence TMPST: Participants received a single dose of ITF2357 100 mg (Treatment T) oral suspension under fasted condition in Period 1, followed by a single dose of moxifloxacin hydrochloride 400 mg tablets (Treatment M) under fasted conditions in Period 2, followed by a single dose of placebo matched to ITL2357 (Treatment P) oral suspension under fasted conditions in Period 3, followed by a single dose of ITF2357 300 mg (as 10 mg/mL, Treatment ST) oral suspension under fasted conditions in Period 4 on Day 1 in the treatment period. Each period was separated by a washout period of 7 days.
- Sequence STPMT: Participants received a single dose of ITF2357 300 mg (as 10 mg/mL, Treatment ST) oral suspension under fasted conditions in Period 1, followed by a single dose of placebo matched to ITL2357 (Treatment P) oral suspension under fasted conditions in Period 2, followed by a single dose of moxifloxacin hydrochloride 400 mg tablets (Treatment M) under fasted conditions in Period 3, followed by a single dose of ITF2357 100 mg (Treatment T) oral suspension under the fasted condition in Period 4 on Day 1 in the treatment period. Each period was separated by a washout period of 7 days.
- Sequence MSTTP: Participants received a single dose of moxifloxacin hydrochloride 400 mg tablets (Treatment M) under fasted conditions in Period 1, followed by a single dose of ITF2357 300 mg (as 10 mg/mL, Treatment ST) oral suspension under fasted conditions in Period 2, followed by a single dose of ITF2357 100 mg (Treatment T) oral suspension under fasted condition in Period 3, followed by a single dose of placebo matched to ITL2357 (Treatment P) oral suspension under fasted conditions in Period 4 on Day 1 in the treatment period. Each period was separated by a washout period of 7 days.
Period: Period 1 (1 Day)
Arm/Group | Sequence TSTPM | Sequence STMTP | Sequence PTMST | Sequence MPSTT | Sequence STPTM | Sequence PMSTT | Sequence TSTMP | Sequence MTPST | Sequence PTSTM | Sequence TMPST | Sequence STPMT | Sequence MSTTP
Started | 1 | 1 | 2 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3
Completed | 1 | 1 | 2 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout Period (7 Days )
Arm/Group | Sequence TSTPM | Sequence STMTP | Sequence PTMST | Sequence MPSTT | Sequence STPTM | Sequence PMSTT | Sequence TSTMP | Sequence MTPST | Sequence PTSTM | Sequence TMPST | Sequence STPMT | Sequence MSTTP
Started | 1 | 1 | 2 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3
Completed | 1 | 1 | 2 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 2 (1 Day)
Arm/Group | Sequence TSTPM | Sequence STMTP | Sequence PTMST | Sequence MPSTT | Sequence STPTM | Sequence PMSTT | Sequence TSTMP | Sequence MTPST | Sequence PTSTM | Sequence TMPST | Sequence STPMT | Sequence MSTTP
Started | 1 | 1 | 2 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3
Completed | 1 | 1 | 2 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout Period (7 Days)
Arm/Group | Sequence TSTPM | Sequence STMTP | Sequence PTMST | Sequence MPSTT | Sequence STPTM | Sequence PMSTT | Sequence TSTMP | Sequence MTPST | Sequence PTSTM | Sequence TMPST | Sequence STPMT | Sequence MSTTP
Started | 1 | 1 | 2 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3
Completed | 1 | 1 | 2 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 3 (1 Day)
Arm/Group | Sequence TSTPM | Sequence STMTP | Sequence PTMST | Sequence MPSTT | Sequence STPTM | Sequence PMSTT | Sequence TSTMP | Sequence MTPST | Sequence PTSTM | Sequence TMPST | Sequence STPMT | Sequence MSTTP
Started | 1 | 1 | 2 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3
Completed | 1 | 1 | 2 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout Period 3 (7 Days)
Arm/Group | Sequence TSTPM | Sequence STMTP | Sequence PTMST | Sequence MPSTT | Sequence STPTM | Sequence PMSTT | Sequence TSTMP | Sequence MTPST | Sequence PTSTM | Sequence TMPST | Sequence STPMT | Sequence MSTTP
Started | 1 | 1 | 2 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3
Completed | 1 | 1 | 2 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 4 (1 Day)
Arm/Group | Sequence TSTPM | Sequence STMTP | Sequence PTMST | Sequence MPSTT | Sequence STPTM | Sequence PMSTT | Sequence TSTMP | Sequence MTPST | Sequence PTSTM | Sequence TMPST | Sequence STPMT | Sequence MSTTP
Started | 1 | 1 | 2 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3
Completed | 1 | 1 | 2 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety population included all participants who had received at least 1 dose of study drug (therapeutic and supratherapeutic doses of ITF2357, moxifloxacin, or placebo). All participants had multiple movement within the arms of the study at different levels and unique participants baseline was not analyzed, only overall participant data was planned, analyzed and reported to avoid double-counting.
Groups:
- All Participants: All participants received a single dose of placebo matched to ITL2357 and moxifloxacin hydrochloride 400 mg tablets under fasted conditions, followed by a single dose of ITF2357 100 and 300 mg oral suspensions in respective 12 fixed sequences (TSTPM, STMTP, PTMST, MPSTT, STPTM, PMSTT, TSTMP, MTPST, PTSTM, TMPST, STPMT, MSTTP) in Periods 1, 2, 3 and 4. Each period was separated by a washout period of 7 days.
Arm/Group | All Participants
Number analyzed (Participants) | 31
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.6 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10
  Not Hispanic or Latino | 21
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 27
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Placebo-corrected Change From Baseline in Fridericia's Corrected QT Interval (QTcF)
Description: The cardio-dynamic assessment was performed through 12-lead electrocardiogram (ECG) extracted from continuous recordings at pre-specified time points. Participants rested in supine position for at least 10 minutes prior to and 5 minutes after each time point for ECG extractions. The QT interval is the time from electrocardiogram Q wave to the end of the T wave corresponding to electrical systole. QT interval was corrected for heart rate using QTcF. Placebo-corrected change from baseline in QTcF (ΔΔQTcF) was calculated based on model-predicted effect.
Time Frame: At 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 7, 8, 12, 24, and 36 hours post-dose
Population: The QT/QTc Population was defined as all participants in the safety population with measurements at baseline as well as on-treatment with at least one post-dose time point with a valid ΔQTcF value. Here, "Overall Number of Participants Analyzed" signifies participants evaluable for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: Milliseconds (msec)
Groups:
- Therapeutic Dose: ITF2357 100 mg: Participants received orally a single dose of ITF2357 100 milligrams (mg; 10 mg per milliliter [mL]) oral suspension and placebo (matched to ITF2357) oral suspension under fasted conditions on Day 1 of Treatment T in each treatment sequence under each assigned period. Each of the 4 periods were separated by a washout of 7 days.
- Supratherapeutic Dose: ITF2357 300 mg: Participants received orally a single dose of ITF2357 300 mg (as 10 mg/mL) oral suspension under fasted conditions on Day 1 of Treatment ST in each treatment sequence under each assigned period. Each of the 4 periods were separated by a washout of 7 days.
- Moxifloxacin: Participants received orally a single dose of moxifloxacin hydrochloride 400 mg tablets under fasted conditions on Day 1 of Treatment M in each treatment sequence under each assigned period. Each of the 4 periods were separated by a washout of 7 days.
Arm/Group | Therapeutic Dose: ITF2357 100 mg | Supratherapeutic Dose: ITF2357 300 mg | Moxifloxacin
Number analyzed (Participants) | 29 | 31 | 30
Milliseconds (msec)
  0.5 hours post-dose | 1.0 (1.06) | 0.5 (1.04) | 10.2 (1.05)
  1 hours post-dose | 0.3 (1.01) | 0.8 (0.99) | 13.1 (1.00)
  1.5 hours Post-dose | 1.0 (0.99) | 2.7 (0.97) | 12.3 (0.98)
  2 hours Post-dose | 2.1 (1.00) | 4.3 (0.98) | 14.0 (0.99)
  2.5 hours Post-dose | 3.6 (1.17) | 6.1 (1.15) | 14.8 (1.16)
  3 hours Post-dose | 2.3 (1.06) | 6.6 (1.04) | 14.0 (1.05)
  3.5 hours Post-dose | 2.8 (1.14) | 9.1 (1.12) | 12.8 (1.13)
  4 hours Post-dose | 4.0 (1.13) | 10.4 (1.11) | 11.9 (1.12)
  5 hours Post-dose | 5.5 (2.11) | 13.6 (2.08) | 12.1 (2.09)
  6 hours Post-dose | 3.8 (1.82) | 11.4 (1.79) | 9.7 (1.81)
  7 hours Post-dose | 3.0 (1.76) | 9.2 (1.73) | 9.6 (1.74)
  8 hours Post-dose | 3.5 (1.57) | 11.5 (1.54) | 11.3 (1.55)
  12 hours Post-dose | 2.5 (1.85) | 10.2 (1.82) | 7.9 (1.83)
  24 hours Post-dose | 2.3 (1.62) | 11.0 (1.59) | 5.6 (1.61)
  36 hours Post-dose | -0.9 (1.86) | 1.5 (1.83) | 1.8 (1.84)

2. Secondary Outcome: Change From Baseline in QTcF Interval
Description: The cardio-dynamic assessment was performed through 12-lead ECGs extracted from continuous recordings at pre-specified time points. Participants rested in supine position for at least 10 minutes prior to and 5 minutes after each time point for ECG extractions. QT interval was corrected for heart rate using Fridericia's correction (QTcF).
Time Frame: At 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 7, 8, 12, 24, and 36 hours post-dose
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: msec
Groups:
- Placebo: Participants received orally a single dose of placebo (matched to ITL2357) oral suspension under fasted conditions on Day 1 of Treatment P in each treatment sequence under each assigned period. Each of the 4 periods were separated by a washout of 7 days.
Arm/Group | Therapeutic Dose: ITF2357 100 mg | Supratherapeutic Dose: ITF2357 300 mg | Moxifloxacin | Placebo
Number analyzed (Participants) | 29 | 31 | 30 | 31
msec
  0.5 hours Post-dose | -0.7 (0.88) | -1.3 (0.86) | 8.5 (0.87) | -1.8 (0.86)
  1 hours Post-dose | -0.3 (0.85) | 0.2 (0.83) | 12.5 (0.84) | -0.6 (0.83)
  1.5 hours Post-dose | 0.8 (0.84) | 2.5 (0.81) | 12.1 (0.82) | -0.2 (0.81)
  2 hours Post-dose | 1.3 (0.85) | 3.6 (0.82) | 13.2 (0.83) | -0.8 (0.82)
  2.5 hours Post-dose | 3.1 (0.95) | 5.5 (0.93) | 14.2 (0.94) | -0.5 (0.93)
  3 hours Post-dose | 2.9 (0.88) | 7.1 (0.86) | 14.5 (0.87) | 0.5 (0.86)
  3.5 hours Post-dose | 4.5 (0.93) | 10.7 (0.91) | 14.4 (0.92) | 1.6 (0.91)
  4 hours Post-dose | 6.0 (0.93) | 12.4 (0.90) | 13.9 (0.91) | 2.0 (0.90)
  5 hours Post-dose | 4.0 (1.58) | 12.1 (1.53) | 10.6 (1.56) | -1.5 (1.53)
  6 hours Post-dose | 0.4 (1.38) | 8.1 (1.34) | 6.3 (1.36) | -3.3 (1.34)
  7 hours Post-dose | -2.3 (1.34) | 3.8 (1.30) | 4.3 (1.32) | -5.3 (1.30)
  8 hours Post-dose | -2.8 (1.21) | 5.2 (1.18) | 5.0 (1.19) | -6.3 (1.18)
  12 hours Post-dose | 3.5 (1.40) | 11.2 (1.36) | 8.8 (1.38) | 1.0 (1.36)
  24 hours Post-dose | -1.5 (1.25) | 7.1 (1.21) | 1.7 (1.23) | -3.9 (1.21)
  36 hours Post-dose | -2.1 (1.41) | 0.2 (1.36) | 0.5 (1.38) | -1.3 (1.36)

3. Secondary Outcome: Change From Baseline in PR Interval
Description: The cardio-dynamic assessment was performed through 12-lead ECGs extracted from continuous recordings at pre-specified time points. Participants rested in supine position for at least 10 minutes prior to and 5 minutes after each time point for ECG extractions. The PR interval is the time from the onset of the P-wave to the start of the next QRS complex, corresponding to the end of atrial depolarization and onset of ventricular depolarization.
Time Frame: At 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 7, 8, 12, 24, and 36 hours post-dose
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: msec
Arm/Group | Therapeutic Dose: ITF2357 100 mg | Supratherapeutic Dose: ITF2357 300 mg | Moxifloxacin | Placebo
Number analyzed (Participants) | 29 | 31 | 30 | 31
msec
  0.5 hours Post-dose | 0.0 (0.83) | -0.7 (0.81) | 0.1 (0.82) | 0.2 (0.81)
  1 hours Post-dose | 0.4 (1.04) | 0.7 (1.01) | -0.3 (1.02) | 2.3 (1.01)
  1.5 hours Post-dose | -1.4 (1.03) | -0.3 (1.00) | -0.4 (1.01) | 1.1 (1.00)
  2 hours Post-dose | 0.4 (1.04) | -1.3 (1.01) | -0.1 (1.02) | 1.6 (1.01)
  2.5 hours Post-dose | -2.4 (1.03) | -2.3 (1.00) | 0.8 (1.00) | -1.9 (1.01)
  3 hours Post-dose | -1.3 (1.03) | -1.6 (1.00) | -1.3 (1.01) | 0.2 (1.00)
  3.5 hours Post-dose | -2.6 (0.97) | -2.8 (0.94) | -2.0 (0.95) | 0.1 (0.94)
  4 hours Post-dose | -2.2 (1.04) | -3.4 (1.01) | -2.6 (1.03) | 0.1 (1.01)
  5 hours Post-dose | -5.3 (1.20) | -7.3 (1.16) | -6.0 (1.18) | -3.2 (1.16)
  6 hours Post-dose | -7.4 (1.30) | -9.3 (1.26) | -8.2 (1.28) | -5.5 (1.26)
  7 hours Post-dose | -7.2 (1.30) | -9.8 (1.26) | -8.0 (1.28) | -5.5 (1.26)
  8 hours Post-dose | -7.4 (1.16) | -9.0 (1.13) | -7.5 (1.15) | -5.2 (1.13)
  12 hours Post-dose | -5.8 (1.39) | -7.9 (1.35) | -6.7 (1.37) | -3.1 (1.35)
  24 hours Post-dose | -3.7 (1.32) | -3.8 (1.28) | 2.1 (1.30) | -0.9 (1.28)
  36 hours Post-dose | -7.8 (1.39) | -9.3 (1.34) | -3.3 (1.36) | -2.6 (1.34)

4. Secondary Outcome: Change From Baseline in QRS Interval
Description: The cardio-dynamic assessment was performed through 12-lead ECGs extracted from continuous recordings at pre-specified time points. Participants rested in supine position for at least 10 minutes prior to and 5 minutes after each time point for ECG extractions. QRS interval is the time from electrocardiogram Q wave to the end of the S wave, corresponding to ventricle depolarization.
Time Frame: At 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 7, 8, 12, 24, and 36 hours post-dose
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: msec
Arm/Group | Therapeutic Dose: ITF2357 100 mg | Supratherapeutic Dose: ITF2357 300 mg | Moxifloxacin | Placebo
Number analyzed (Participants) | 29 | 31 | 30 | 31
msec
  0.5 hours Post-dose | -0.1 (0.14) | 0.1 (0.13) | 0.2 (0.14) | 0.2 (0.13)
  1 hours Post-dose | 0.2 (0.16) | 0.1 (0.16) | 0.4 (0.16) | 0.0 (0.16)
  1.5 hours Post-dose | 0.0 (0.16) | 0.0 (0.16) | -0.1 (0.16) | -0.1 (0.16)
  2 hours Post-dose | -0.1 (0.15) | 0.2 (0.15) | 0.2 (0.15) | 0.0 (0.15)
  2.5 hours Post-dose | -0.1 (0.17) | 0.2 (0.16) | 0.3 (0.16) | 0.1 (0.16)
  3 hours Post-dose | 0.1 (0.17) | 0.4 (0.17) | 0.3 (0.17) | 0.3 (0.17)
  3.5 hours Post-dose | 0.1 (0.18) | 0.5 (0.17) | 0.1 (0.18) | 0.3 (0.17)
  4 hours Post-dose | 0.1 (0.20) | 0.4 (0.19) | 0.3 (0.20) | 0.2 (0.19)
  5 hours Post-dose | 0.1 (0.27) | 0.5 (0.26) | 0.3 (0.27) | 0.5 (0.26)
  6 hours Post-dose | -0.4 (0.24) | -0.3 (0.24) | -0.4 (0.24) | -0.2 (0.24)
  7 hours Post-dose | -0.7 (0.24) | -0.6 (0.23) | -0.5 (0.23) | -0.2 (0.23)
  8 hours Post-dose | -0.5 (0.22) | 0.1 (0.21) | -0.2 (0.21) | -0.2 (0.21)
  12 hours Post-dose | 0.2 (0.30) | -0.2 (0.29) | 0.1 (0.29) | 0.3 (0.29)
  24 hours Post-dose | -0.3 (0.39) | 0.1 (0.38) | -0.5 (0.39) | -0.3 (0.38)
  36 hours Post-dose | -0.4 (0.27) | -0.4 (0.26) | -0.5 (0.26) | -0.3 (0.26)

5. Secondary Outcome: Change From Baseline in Heart Rate (HR) Interval
Description: The cardio-dynamic assessment was performed through 12-lead ECGs extracted from continuous recordings at pre-specified time points. Participants rested in supine position for at least 10 minutes prior to and 5 minutes after each time point for ECG extractions. Baseline is defined as the last results (scheduled or unscheduled) obtained prior to drug administration in each period.
Time Frame: At 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 7, 8, 12, 24, and 36 hours post-dose
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: beats per minute (bpm)
Arm/Group | Therapeutic Dose: ITF2357 100 mg | Supratherapeutic Dose: ITF2357 300 mg | Moxifloxacin | Placebo
Number analyzed (Participants) | 29 | 31 | 30 | 31
beats per minute (bpm)
  0.5 hours Post-dose | 0.6 (0.76) | 1.1 (0.75) | 1.3 (0.75) | 0.5 (0.75)
  1 hours Post-dose | 1.2 (0.85) | 2.8 (0.83) | 2.3 (0.84) | 1.1 (0.83)
  1.5 hours Post-dose | 3.3 (0.85) | 5.1 (0.83) | 1.9 (0.84) | 1.1 (0.84)
  2 hours Post-dose | 3.7 (0.86) | 7.8 (0.84) | 1.4 (0.85) | 1.1 (0.84)
  2.5 hours Post-dose | 3.8 (0.99) | 9.9 (0.97) | 0.9 (0.98) | 0.5 (0.97)
  3 hours Post-dose | 4.3 (0.86) | 10.5 (0.84) | 1.4 (0.85) | 0.7 (0.84)
  3.5 hours Post-dose | 4.0 (0.89) | 9.9 (0.87) | 2.2 (0.88) | 0.1 (0.87)
  4 hours Post-dose | 4.3 (0.94) | 11.0 (0.92) | 2.3 (0.93) | 1.3 (0.92)
  5 hours Post-dose | 15.0 (1.00) | 22.1 (0.98) | 10.6 (0.99) | 10.5 (0.98)
  6 hours Post-dose | 12.4 (1.10) | 21.7 (1.07) | 10.2 (1.08) | 10.4 (1.07)
  7 hours Post-dose | 8.2 (1.04) | 17.0 (1.02) | 7.5 (1.03) | 6.7 (1.02)
  8 hours Post-dose | 7.4 (0.88) | 14.0 (0.86) | 6.2 (0.87) | 5.6 (0.86)
  12 hours Post-dose | 9.5 (1.14) | 12.7 (1.11) | 10.6 (1.13) | 10.6 (1.11)
  24 hours Post-dose | 0.6 (0.80) | 2.1 (0.79) | 1.6 (0.80) | 2.2 (0.79)
  36 hours Post-dose | 9.1 (1.18) | 8.1 (1.15) | 10.2 (1.16) | 9.9 (1.15)

6. Secondary Outcome: Placebo-corrected Change From Baseline in PR Interval
Description: Placebo-corrected change from Baseline in PR, (ΔΔPR) was calculated based on model-predicted effect. PR interval was the time between the beginning of the P wave and the start of the QRS interval, corresponding to the end of atrial depolarization and onset of ventricular depolarization.
Time Frame: At 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 7, 8, 12, 24, and 36 hours post-dose
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: msec
Arm/Group | Therapeutic Dose: ITF2357 100 mg | Supratherapeutic Dose: ITF2357 300 mg | Moxifloxacin
Number analyzed (Participants) | 29 | 31 | 30
msec
  0.5 hours Post-dose | -0.2 (1.02) | -0.9 (1.00) | -0.1 (1.01)
  1 hour Post-dose | -1.9 (1.34) | -1.6 (1.31) | -2.6 (1.32)
  1.5 hours Post-dose | -2.6 (1.33) | -1.5 (1.30) | -1.6 (1.31)
  2 hours Post-dose | -1.2 (1.34) | -2.9 (1.31) | -1.7 (1.32)
  2.5 hours Post-dose | -3.2 (1.32) | -3.1 (1.30) | -2.6 (1.31)
  3 hour Post-dose | -1.4 (1.32) | -1.8 (1.30) | -1.5 (1.31)
  3.5 hours Post-dose | -2.7 (1.23) | -2.9 (1.21) | -2.1 (1.22)
  4 hours Post-dose | -2.3 (1.35) | -3.5 (1.32) | -2.6 (1.33)
  5 hours Post-dose | -2.1 (1.57) | -4.1 (1.55) | -2.8 (1.56)
  6 hours Post-dose | -1.9 (1.73) | -3.8 (1.70) | -2.7 (1.71)
  7 hours Post-dose | -1.7 (1.73) | -4.3 (1.70) | -2.5 (1.71)
  8 hours Post-dose | -2.2 (1.53) | -3.8 (1.50) | -2.3 (1.51)
  12 hours Post-dose | -2.7 (1.85) | -4.7 (1.82) | -3.6 (1.84)
  24 hours Post-dose | -2.8 (1.76) | -2.9 (1.73) | 3.0 (1.74)
  36 hours Post-dose | -5.2 (1.85) | -6.6 (1.82) | -0.7 (1.83)

7. Secondary Outcome: Placebo-corrected Change From Baseline in QRS Interval
Description: Placebo-corrected change from baseline for QRS interval, (ΔΔQRS) was calculated based on model-predicted effect. QRS interval is the time from Q wave to the end of the S wave, corresponding to ventricle depolarization.
Time Frame: At 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 7, 8, 12, 24, and 36 hours post-dose
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: msec
Arm/Group | Therapeutic Dose: ITF2357 100 mg | Supratherapeutic Dose: ITF2357 300 mg | Moxifloxacin
Number analyzed (Participants) | 29 | 31 | 30
msec
  0.5 hours Post-dose | -0.2 (0.17) | 0.0 (0.16) | 0.1 (0.17)
  1 hours Post-dose | 0.1 (0.21) | 0.1 (0.20) | 0.4 (0.20)
  1.5 hours Post-dose | 0.1 (0.21) | 0.1 (0.20) | 0.0 (0.20)
  2 hours Post-dose | 0.0 (0.19) | 0.2 (0.19) | 0.3 (0.19)
  2.5 hours Post-dose | -0.2 (0.21) | 0.1 (0.20) | 0.2 (0.21)
  3 hours Post-dose | -0.2 (0.22) | 0.1 (0.22) | 0.0 (0.22)
  3.5 hours Post-dose | -0.3 (0.23) | 0.2 (0.23) | -0.2 (0.23)
  4 hours Post-dose | 0.0 (0.26) | 0.2 (0.26) | 0.2 (0.26)
  5 hours Post-dose | -0.3 (0.37) | 0.0 (0.36) | -0.2 (0.36)
  6 hours Post-dose | -0.2 (0.32) | 0.0 (0.32) | -0.1 (0.32)
  7 hours Post-dose | -0.5 (0.32) | -0.4 (0.31) | -0.3 (0.31)
  8 hours Post-dose | -0.3 (0.28) | 0.2 (0.28) | 0.0 (0.28)
  12 hours Post-dose | 0.0 (0.40) | -0.5 (0.39) | -0.1 (0.40)
  24 hours Post-dose | 0.1 (0.54) | 0.4 (0.53) | -0.1 (0.53)
  36 hours Post-dose | -0.1 (0.36) | -0.1 (0.35) | -0.2 (0.36)

8. Secondary Outcome: Placebo-corrected Change From Baseline in HR Interval
Description: Placebo-corrected change from baseline in HR, (ΔΔHR) was calculated based on model-predicted effect.
Time Frame: At 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 7, 8, 12, 24, and 36 hours post-dose
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: bpm
Arm/Group | Therapeutic Dose: ITF2357 100 mg | Supratherapeutic Dose: ITF2357 300 mg | Moxifloxacin
Number analyzed (Participants) | 29 | 31 | 30
bpm
  0.5 hours Post-dose | 0.1 (0.73) | 0.6 (0.71) | 0.8 (0.72)
  1 hours Post-dose | 0.1 (0.89) | 1.6 (0.88) | 1.2 (0.88)
  1.5 hours Post-dose | 2.2 (0.90) | 4.0 (0.88) | 0.8 (0.89)
  2 hours Post-dose | 2.6 (0.92) | 6.7 (0.90) | 0.3 (0.91)
  2.5 hours Post-dose | 3.3 (1.15) | 9.3 (1.13) | 0.3 (1.14)
  3 hours Post-dose | 3.6 (0.91) | 9.8 (0.90) | 0.7 (0.91)
  3.5 hours Post-dose | 3.9 (0.96) | 9.8 (0.95) | 2.1 (0.96)
  4 hours Post-dose | 3.0 (1.06) | 9.7 (1.04) | 1.0 (1.05)
  5 hours Post-dose | 4.5 (1.17) | 11.6 (1.15) | 0.1 (1.16)
  6 hours Post-dose | 1.9 (1.32) | 11.2 (1.29) | -0.3 (1.31)
  7 hours Post-dose | 1.4 (1.23) | 10.2 (1.21) | 0.7 (1.22)
  8 hours Post-dose | 1.9 (0.95) | 8.5 (0.93) | 0.7 (0.94)
  12 hours Post-dose | -1.1 (1.39) | 2.1 (1.37) | -0.1 (1.38)
  24 hours Post-dose | -1.6 (0.82) | -0.2 (0.80) | -0.7 (0.81)
  36 hours Post-dose | -0.8 (1.45) | -1.8 (1.43) | 0.3 (1.44)

9. Secondary Outcome: Number of Participants With Changes in Categorical Outliers for QTcF, PR, and QRS Intervals in the ECG and HR
Description: QTcF:
  Treatment-emergent value of greater than (>) 450 and less than or equal to (<=) 480 ms when not present at Baseline (new onset).
  Treatment-emergent value of > 480 and <= 500 ms when not present at Baseline (new onset).
  Treatment-emergent value of > 500 ms when not present at Baseline (new onset). Increase of QTcF (ΔQTcF) from Baseline of > 30 and <= 60 ms. Increase of QTcF from Baseline > 60 ms
  HR:
  Decrease of HR from Baseline > 25% resulting in HR less than (<) 50 bpm. Increase of HR from Baseline > 25% resulting in HR > 100 bpm.
  PR:
  Increase of PR from Baseline > 25% resulting in PR > 210 ms.
  QRS:
  Increase of QRS from Baseline > 25% resulting in QRS > 120 ms.
Time Frame: Baseline, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 7, 8, 12, 24, and 36 hours post-dose
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Therapeutic Dose: ITF2357 100 mg | Supratherapeutic Dose: ITF2357 300 mg | Moxifloxacin | Placebo
Number analyzed (Participants) | 29 | 31 | 30 | 31
Participants
  QTcF > 450 and <= 480 ms | 0 | 1 | 2 | 0
  QTcF > 480 and <= 500 ms | 0 | 0 | 0 | 0
  QTcF > 500 ms | 0 | 0 | 0 | 0
  ΔQTcF > 30 and <= 60 ms | 0 | 2 | 2 | 0
  ΔQTcF > 60 ms | 0 | 0 | 0 | 0
  HR < 50 (bpm) with a decrease in ΔHR > 25% | 0 | 0 | 0 | 0
  HR > 100 (bpm) with an increase in ΔHR > 25% | 0 | 0 | 0 | 0
  PR > 210 (ms) with an increase in ΔPR > 25% | 0 | 0 | 0 | 0
  QRS > 120 (ms) with an increase in ΔQRS > 25% | 0 | 0 | 0 | 0

10. Secondary Outcome: Number of Participants With Treatment-Emergent Changes of T-Wave Morphology and U Wave Presence
Description: T-wave abnormalities were categorized as follows:
  Normal T wave (+): Any positive T wave not meeting any criterion below. Flat T wave: T amplitude < 1 mm (either positive or negative) including flat isoelectric line.
  Notched T wave (+): Presence of notch(es) of at least 0.05 mV amplitude on ascending or descending arm of the positive T wave.
  Biphasic: T wave that contains a second component with an opposite phase that is at least 0.1 mV deep (both positive/negative and negative/positive and polyphasic T waves included).
  Normal T wave (-): T amplitude that is negative, without biphasic T wave or notches.
  Notched T wave (-): Presence of notch(es) of at least 0.05 mV amplitude on descending or ascending arm of the negative T wave.
  U waves: Presence of abnormal U waves.
Time Frame: Up to 44 days
Population: The safety population was defined as all participants who received at least 1 dose of study drug (therapeutic and supratherapeutic doses of ITF2357, moxifloxacin, or placebo). Here, "Overall Number of Participants Analyzed" signifies participants evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Therapeutic Dose: ITF2357 100 mg | Supratherapeutic Dose: ITF2357 300 mg | Moxifloxacin | Placebo
Number analyzed (Participants) | 29 | 31 | 30 | 31
Participants
  Flat | 0 | 0 | 0 | 0
  Notched (+) | 0 | 0 | 0 | 0
  Biphasic | 0 | 0 | 0 | 0
  Normal (-) | 0 | 0 | 0 | 0
  Notched (-) | 0 | 0 | 0 | 0
  U-Wave presence | 0 | 0 | 0 | 0

11. Secondary Outcome: Plasma Pharmacokinetic (PK): Area Under the Concentration-Time Curve From Time Zero to the Last Measurable Concentration (AUC0-t) of ITF2357 and Its Metabolites
Description: The area under the concentration time curve (AUC) from time zero (= dosing time) to the last sampling time (tlast) at which the concentration is at or above the lower limit of quantification. AUC0-t was calculated using the mixed log-linear trapezoidal rule (linear up, log down). AUC0-t of ITF2357 and metabolites: ITF2374, ITF2375, ITF2440, ITF2563, and ITF2955 glucuronide were reported.
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 7, 8, 12, 24, 36, 48, 60, and 72 hours post-dose
Population: The PK population was defined as all participants who completed at least 3 periods, including at least Treatments T, ST, and M for whom the PK profile was adequately characterized. Here, "Number Analyzed" signified participants who were evaluable for this outcome measure at specified category.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours*nanograms per milliliter (h*ng/mL)
Arm/Group | Therapeutic Dose: ITF2357 100 mg | Supratherapeutic Dose: ITF2357 300 mg
Number analyzed (Participants) | 29 | 29
hours*nanograms per milliliter (h*ng/mL)
  ITF2357 | 596.10 (22.57) | 2313.44 (20.53)
  ITF2374: number analyzed (Participants) | 12 | 12
  ITF2374 | 363.55 (63.83) | 1296.22 (59.65)
  ITF2375: number analyzed (Participants) | 12 | 12
  ITF2375 | 2672.92 (54.88) | 9599.11 (52.70)
  ITF2440: number analyzed (Participants) | 12 | 12
  ITF2440 | 5696.28 (23.36) | 18577.74 (21.34)
  ITF2563: number analyzed (Participants) | 12 | 12
  ITF2563 | 1247.92 (23.58) | 3563.33 (20.59)
  ITF2955 glucuronide: number analyzed (Participants) | 4 | 12
  ITF2955 glucuronide | 1.53 (78.00) | 15.89 (47.69)

12. Secondary Outcome: Plasma PK: Area Under the Concentration-Time Curve From Time Zero to the Last Measurable Concentration (AUC0-t) of Moxifloxacin
Description: The area under the concentration time curve (AUC) from time zero (= dosing time) to the last sampling time (tlast) at which the concentration is at or above the lower limit of quantification. AUC0-t was calculated using the mixed log-linear trapezoidal rule (linear up, log down).
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 7, 8, 12, 24, 36, 48, 60, and 72 hours post-dose
Population: The PK population was defined as all participants who completed at least 3 periods, including at least Treatments T, ST, and M for whom the PK profile was adequately characterized.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Moxifloxacin
Number analyzed (Participants) | 29
h*ng/mL | 27077.52 (16.17)

13. Secondary Outcome: Plasma PK: Area Under the Concentration-Time Curve From Time Zero to 12 Hours (AUC0-12) of ITF2357 and Its Metabolites
Description: AUC0-12 was calculated using the trapezoidal method for ITF2357 and metabolites: ITF2374, ITF2375, ITF2440, ITF2563, and ITF2955 glucuronide. AUC0-12:: of ITF2357 and its metabolites: ITF2374, ITF2375, ITF2440, ITF2563, and ITF2955 glucuronide were reported.
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 7, 8, and 12 hours post-dose
Population: The PK population was defined as all participants who completed at least 3 periods, including at least Treatments T, ST, and M for whom the PK profile was adequately characterized. Here, "Number Analyzed" signifies participants who were evaluable for this outcome measure at specified category.
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Therapeutic Dose: ITF2357 100 mg | Supratherapeutic Dose: ITF2357 300 mg
Number analyzed (Participants) | 29 | 29
h*ng/mL
  ITF2357 | 480.70 (114.09) | 1893.60 (423.33)
  ITF2374: number analyzed (Participants) | 12 | 12
  ITF2374 | 178.10 (81.57) | 607.16 (258.73)
  ITF2375: number analyzed (Participants) | 12 | 12
  ITF2375 | 1680.76 (725.80) | 6018.02 (2430.06)
  ITF2440: number analyzed (Participants) | 12 | 12
  ITF2440 | 1448.97 (362.63) | 3924.21 (1130.05)
  ITF2563: number analyzed (Participants) | 12 | 12
  ITF2563 | 299.77 (85.39) | 776.22 (259.98)
  ITF2955 glucuronide: number analyzed (Participants) | 12 | 12
  ITF2955 glucuronide | 0.88 (1.62) | 18.08 (8.39)

14. Secondary Outcome: Plasma PK: Area Under the Concentration-Time Curve From Time Zero to 12 Hours (AUC0-12) of Moxifloxacin
Description: AUC0-12 was calculated using the trapezoidal method for Moxifloxacin.
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 7, 8 and 12 hours post-dose
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Moxifloxacin
Number analyzed (Participants) | 29
h*ng/mL | 13625.09 (2733.45)

15. Secondary Outcome: Plasma PK: Area Under the Concentration-Time Curve From Time Zero to Infinity (AUC0-inf) of ITF2357 and Its Metabolites
Description: AUC0-inf was calculated as AUC0-t + Clast/Kel, where Clast is the last measurable concentration. Elimination rate constant (Kel),was defined as the negative of the estimated slope of the linear regression of the in-transformed concentration versus time profile in the terminal elimination phase. AUC0-inf of ITF2357 and metabolites: ITF2374, ITF2375, ITF2440, ITF2563, and ITF2955 glucuronide were reported.
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 7, 8, 12, 24, 36, 48, 60, and 72 hours post-dose
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Therapeutic Dose: ITF2357 100 mg | Supratherapeutic Dose: ITF2357 300 mg
Number analyzed (Participants) | 29 | 29
h*ng/mL
  ITF2357 | 626.57 (139.54) | 2383.27 (484.72)
  ITF2374: number analyzed (Participants) | 12 | 12
  ITF2374 | 475.82 (318.25) | 1555.70 (986.40)
  ITF2375: number analyzed (Participants) | 12 | 12
  ITF2375 | 3246.97 (1806.52) | 11373.93 (6045.30)
  ITF2440: number analyzed (Participants) | 12 | 12
  ITF2440 | 6196.74 (1400.60) | 19920.16 (4134.67)
  ITF2563: number analyzed (Participants) | 12 | 12
  ITF2563 | 1357.46 (290.51) | 3864.88 (757.94)
  ITF2955 glucuronide: number analyzed (Participants) | 1 | 9
  ITF2955 glucuronide | 10.20 | 20.68 (9.56)

16. Secondary Outcome: Plasma PK: Area Under the Concentration-Time Curve From Time Zero to Infinity (AUC0-inf) of Moxifloxacin
Description: AUC0-inf was calculated as AUC0-t + Clast/Kel, where Clast is the last measurable concentration for Moxifloxacin.
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 7, 8, 12, 24, 36, 48, 60, and 72 hours post-dose
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Moxifloxacin
Number analyzed (Participants) | 29
h*ng/mL | 28327.15 (4616.50)

17. Secondary Outcome: Plasma PK: Percentage of Residual Area for ITF2357 and Its Metabolites
Description: Residual area was calculated as 100*(1- AUC0-t / AUC0-inf) for ITF2357 and Metabolites: ITF2374, ITF2375, ITF2440, ITF2563, and ITF2955 glucuronide.
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 7, 8, 12, 24, 36, 48, 60, and 72 hours post-dose
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: Percentage of residual area
Arm/Group | Therapeutic Dose: ITF2357 100 mg | Supratherapeutic Dose: ITF2357 300 mg
Number analyzed (Participants) | 29 | 29
Percentage of residual area
  ITF2357 | 2.63 (0.84) | 0.95 (0.36)
  ITF2374: number analyzed (Participants) | 12 | 12
  ITF2374 | 8.49 (4.23) | 3.72 (2.82)
  ITF2375: number analyzed (Participants) | 12 | 12
  ITF2375 | 3.45 (2.28) | 1.70 (1.25)
  ITF2440: number analyzed (Participants) | 12 | 12
  ITF2440 | 5.81 (3.09) | 4.69 (3.58)
  ITF2563: number analyzed (Participants) | 12 | 12
  ITF2563 | 6.04 (4.53) | 5.95 (4.42)
  ITF2955 glucuronide: number analyzed (Participants) | 1 | 9
  ITF2955 glucuronide | 66.07 | 24.01 (6.03)

18. Secondary Outcome: Plasma PK: Percentage of Residual Area for Moxifloxacin
Description: Residual area was calculated as 100*(1- AUC0-t / AUC0-inf) for moxifloxacin.
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 7, 8, 12, 24, 36, 48, 60, and 72 hours post-dose
Population: as for outcome 12
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Percentage of residual area
Arm/Group | Moxifloxacin
Number analyzed (Participants) | 29
Percentage of residual area | 2.81 (48.66)

19. Secondary Outcome: Plasma PK: Maximum Observed Plasma Concentration (Cmax) of ITF2357 and Its Metabolites
Description: Cmax was calculated for ITF2357 and Metabolites: ITF2374, ITF2375, ITF2440, ITF2563, and ITF2955 glucuronide. Cmax was taken directly from the observed concentration-time curve.
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 7, 8, 12, 24, 36, 48, 60, and 72 hours post-dose
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Therapeutic Dose: ITF2357 100 mg | Supratherapeutic Dose: ITF2357 300 mg
Number analyzed (Participants) | 29 | 29
ng/mL
  ITF2357 | 102.84 (30.55) | 409.65 (133.74)
  ITF2374: number analyzed (Participants) | 12 | 12
  ITF2374 | 24.39 (11.01) | 81.59 (32.93)
  ITF2375: number analyzed (Participants) | 12 | 12
  ITF2375 | 258.64 (111.23) | 820.75 (273.52)
  ITF2440: number analyzed (Participants) | 12 | 12
  ITF2440 | 195.23 (45.41) | 602.02 (142.15)
  ITF2563: number analyzed (Participants) | 12 | 12
  ITF2563 | 43.90 (13.03) | 123.27 (31.02)
  ITF2955 glucuronide: number analyzed (Participants) | 12 | 12
  ITF2955 glucuronide | 0.42 (0.62) | 4.41 (1.70)

20. Secondary Outcome: Plasma PK: Maximum Observed Plasma Concentration (Cmax) of Moxifloxacin
Description: Cmax was calculated for moxifloxacin. Cmax was taken directly from the observed concentration-time curve.
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 7, 8, 12, 24, 36, 48, 60, and 72 hours post-dose
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Moxifloxacin
Number analyzed (Participants) | 29
ng/mL | 1789.49 (498.08)

21. Secondary Outcome: Plasma PK: Time of Observed Cmax (Tmax) of ITF2357 and Its Metabolites
Description: Tmax was calculated for ITF2357 and Metabolites: ITF2374, ITF2375, ITF2440, ITF2563, and ITF2955 glucuronide. The time to reach the maximum observed plasma concentration obtained directly from plasma concentration time curve.
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 7, 8, 12, 24, 36, 48, 60, and 72 hours post-dose
Population: as for outcome 13
Measure: Median (Full Range); unit: hours
Arm/Group | Therapeutic Dose: ITF2357 100 mg | Supratherapeutic Dose: ITF2357 300 mg
Number analyzed (Participants) | 29 | 29
hours
  ITF2357 | 2.139 [1.099 to 3.355] | 2.158 [1.165 to 5.092]
  ITF2374: number analyzed (Participants) | 12 | 12
  ITF2374 | 5.098 [5.089 to 6.298] | 5.634 [5.093 to 7.094]
  ITF2375: number analyzed (Participants) | 12 | 12
  ITF2375 | 3.610 [2.153 to 4.101] | 4.094 [2.599 to 5.101]
  ITF2440: number analyzed (Participants) | 12 | 12
  ITF2440 | 12.144 [8.090 to 12.238] | 12.152 [12.134 to 12.228]
  ITF2563: number analyzed (Participants) | 12 | 29
  ITF2563 | 12.146 [7.100 to 12.238] | 12.152 [8.090 to 12.228]
  ITF2955 glucuronide: number analyzed (Participants) | 12 | 12
  ITF2955 glucuronide | 0 [0 to 3.604] | 2.606 [1.596 to 4.093]

22. Secondary Outcome: Plasma PK: Time of Observed Cmax (Tmax) of Moxifloxacin
Description: Tmax was calculated for Moxifloxacin. The time to reach the maximum observed plasma concentration obtained directly from plasma concentration time curve.
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 7, 8, 12, 24, 36, 48, 60, and 72 hours post-dose
Population: as for outcome 12
Measure: Mean (Full Range); unit: hours
Arm/Group | Moxifloxacin
Number analyzed (Participants) | 29
hours | 2.327 [0.615 to 4.095]

23. Secondary Outcome: Plasma PK: Elimination Rate Constant (Kel) of ITF2357 and Its Metabolites
Description: Kel was defined as the negative of the estimated slope of the linear regression of the ln-transformed concentration versus time profile in the terminal elimination phase. Kel was calculated for ITF2357 and Metabolites: ITF2374, ITF2375, ITF2440, ITF2563, andITF2955 glucuronide.
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 7, 8, 12, 24, 36, 48, 60, and 72 hours post-dose
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: fraction per hour
Arm/Group | Therapeutic Dose: ITF2357 100 mg | Supratherapeutic Dose: ITF2357 300 mg
Number analyzed (Participants) | 29 | 29
fraction per hour
  ITF2357 | 0.0923 (0.0198) | 0.0652 (0.0146)
  ITF2374: number analyzed (Participants) | 12 | 12
  ITF2374 | 0.0570 (0.0141) | 0.0549 (0.0175)
  ITF2375: number analyzed (Participants) | 12 | 12
  ITF2375 | 0.0585 (0.0157) | 0.0667 (0.0130)
  ITF2440: number analyzed (Participants) | 12 | 12
  ITF2440 | 0.0508 (0.0126) | 0.0530 (0.0124)
  ITF2563: number analyzed (Participants) | 12 | 12
  ITF2563 | 0.0499 (0.0138) | 0.0498 (0.0156)
  ITF2955 glucuronide: number analyzed (Participants) | 1 | 9
  ITF2955 glucuronide | 0.1514 | 0.2886 (0.0944)

24. Secondary Outcome: Plasma PK: Elimination Rate Constant (Kel) of Moxifloxacin
Description: Kel was defined as the negative of the estimated slope of the linear regression of the ln-transformed concentration versus time profile in the terminal elimination phase. Kel was calculated for Moxifloxacin.
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 7, 8, 12, 24, 36, 48, 60, and 72 hours post-dose
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: fraction per hour
Arm/Group | Moxifloxacin
Number analyzed (Participants) | 29
fraction per hour | 0.0493 (0.0091)

25. Secondary Outcome: Plasma PK: Elimination Half-life (T½ el) of ITF2357 and Its Metabolites
Description: T½ el was calculated as ln(2)/kel for ITF2357 and Metabolites : ITF2374, ITF2375, ITF2440, ITF2563, ITF2955 glucuronide, and Moxifloxacin.
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 7, 8, 12, 24, 36, 48, 60, and 72 hours post-dose
Population: as for outcome 13
Measure: Median (Full Range); unit: hours
Arm/Group | Therapeutic Dose: ITF2357 100 mg | Supratherapeutic Dose: ITF2357 300 mg
Number analyzed (Participants) | 29 | 29
hours
  ITF2357 | 7.25 [5.47 to 13.69] | 11.19 [6.26 to 16.35]
  ITF2374: number analyzed (Participants) | 12 | 12
  ITF2374 | 12.63 [9.08 to 26.30] | 12.49 [8.27 to 22.07]
  ITF2375: number analyzed (Participants) | 12 | 12
  ITF2375 | 12.31 [8.38 to 16.77] | 10.71 [7.97 to 13.86]
  ITF2440: number analyzed (Participants) | 12 | 12
  ITF2440 | 12.91 [9.94 to 22.65] | 13.07 [9.48 to 20.87]
  ITF2563: number analyzed (Participants) | 12 | 12
  ITF2563 | 13.47 [9.76 to 29.08] | 13.33 [9.56 to 23.00]
  ITF2955 glucuronide: number analyzed (Participants) | 1 | 9
  ITF2955 glucuronide | 4.58 [4.58 to 4.58] | 2.27 [1.62 to 4.49]

26. Secondary Outcome: Plasma PK: Elimination Half-life (T½ el) of Moxifloxacin
Description: T½ el was calculated as ln(2)/kel for moxifloxacin.
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 7, 8, 12, 24, 36, 48, 60, and 72 hours post-dose
Population: as for outcome 12
Measure: Median (Full Range); unit: hours
Arm/Group | Moxifloxacin
Number analyzed (Participants) | 29
hours | 13.97 [9.96 to 20.83]

27. Secondary Outcome: Plasma PK: Apparent Total Body Clearance (CL/F) of ITF2357 and Its Metabolites
Description: CL/F was calculated as Dose/AUC0-inf for ITF2357 and Metabolites: ITF2374, ITF2375, ITF2440, ITF2563, and ITF2955 glucuronide.
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 7, 8, 12, 24, 36, 48, 60, and 72 hours post-dose
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: liters per hour
Arm/Group | Therapeutic Dose: ITF2357 100 mg | Supratherapeutic Dose: ITF2357 300 mg
Number analyzed (Participants) | 29 | 29
liters per hour
  ITF2357 | 167.12 (36.40) | 131.11 (27.51)
  ITF2374: number analyzed (Participants) | 12 | 12
  ITF2374 | 296.86 (172.71) | 251.84 (124.72)
  ITF2375: number analyzed (Participants) | 12 | 12
  ITF2375 | 43.11 (27.80) | 36.69 (23.96)
  ITF2440: number analyzed (Participants) | 12 | 12
  ITF2440 | 16.94 (4.01) | 15.73 (3.60)
  ITF2563: number analyzed (Participants) | 12 | 12
  ITF2563 | 76.77 (16.33) | 80.71 (17.61)
  ITF2955 glucuronide: number analyzed (Participants) | 1 | 9
  ITF2955 glucuronide | 9808.03 | 16631.81 (5576.18)

28. Secondary Outcome: Plasma PK: Apparent Total Body Clearance (CL/F) of Moxifloxacin
Description: CL/F was calculated as Dose/AUC0-inf for moxifloxacin.
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 7, 8, 12, 24, 36, 48, 60, and 72 hours post-dose
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: liters per hour
Arm/Group | Moxifloxacin
Number analyzed (Participants) | 29
liters per hour | 14.49 (2.39)

29. Secondary Outcome: Plasma PK: Apparent Volume of Distribution (Vd/F) of ITF2357 and Its Metabolites
Description: Vd/F was calculated as Dose/Kel x AUC0-inf for ITF2357 and Metabolites: ITF2374, ITF2375, ITF2440, ITF2563, and ITF2955 glucuronide.
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 7, 8, 12, 24, 36, 48, 60, and 72 hours post-dose
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: liters
Arm/Group | Therapeutic Dose: ITF2357 100 mg | Supratherapeutic Dose: ITF2357 300 mg
Number analyzed (Participants) | 29 | 29
liters
  ITF2357 | 1897.03 (588.15) | 2125.49 (764.32)
  ITF2374: number analyzed (Participants) | 12 | 12
  ITF2374 | 5094.92 (2676.37) | 5027.46 (3106.93)
  ITF2375: number analyzed (Participants) | 12 | 12
  ITF2375 | 795.34 (636.25) | 576.42 (436.72)
  ITF2440: number analyzed (Participants) | 12 | 12
  ITF2440 | 354.01 (123.39) | 311.58 (96.04)
  ITF2563: number analyzed (Participants) | 12 | 12
  ITF2563 | 1702.58 (749.67) | 1757.38 (556.98)
  ITF2955 glucuronide: number analyzed (Participants) | 1 | 9
  ITF2955 glucuronide | 64779.37 | 58366.39 (12977.61)

30. Secondary Outcome: Plasma PK: Apparent Volume of Distribution (Vd/F) of Moxifloxacin
Description: Vd/F was calculated as Dose/Kel x AUC0-inf for moxifloxacin.
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 7, 8, 12, 24, 36, 48, 60, and 72 hours post-dose
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: liters
Arm/Group | Moxifloxacin
Number analyzed (Participants) | 29
liters | 303.02 (72.21)

31. Secondary Outcome: Urine PK: Cumulative Urinary Excretion From Time Zero to Time t (Ae0-t) for ITF2357 and Its Metabolites
Description: Ae0-t was calculated as the sum of the amounts excreted over each collection interval. The amount excreted in the urine for each time interval is calculated as the urine concentration multiplied by the urine volume for ITF2357 and Metabolites: ITF2374, ITF2375, ITF2440, ITF2563, ITF2955 glucuronide.
Time Frame: Pre-dose (within 2 hours before dosing), 0-8 hours, 8-24 hours, 24-48 hours, and 48-72 hours post-dose
Population: The PK population was defined as all participants who completed at least 3 periods, including at least Treatments T, ST, and M for whom the PK profile was adequately characterized. Here, "Overall Number of Participants Analyzed" signifies participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Nanograms (ng)
Arm/Group | Therapeutic Dose: ITF2357 100 mg | Supratherapeutic Dose: ITF2357 300 mg
Number analyzed (Participants) | 12 | 12
Nanograms (ng)
  ITF2357 | 1304747.81 (444627.39) | 4284095.88 (1031461.74)
  ITF2374 | 1526630.97 (820295.42) | 4634585.90 (2469826.92)
  ITF2375 | 330005.73 (244198.09) | 1051751.97 (702770.77)
  ITF2440 | 20496643.63 (3002369.96) | 55319154.12 (9058968.83)
  ITF2563 | 9746260.02 (1204246.03) | 27259547.79 (4213356.29)
  ITF2955 glucuronide | 13456.18 (3086.53) | 66582.99 (18731.80)

32. Secondary Outcome: Urine PK: Maximum Rate of Urinary Excretion (Rmax) for ITF2357 and Its Metabolites
Description: Rmax was calculated by dividing the amount of drug excreted in each collection interval by the time over which it was collected for ITF2357 and Metabolites: ITF2374, ITF2375, ITF2440, ITF2563, ITF2955 glucuronide.
Time Frame: Pre-dose (within 2 hours before dosing), 0-8 hours, 8-24 hours, 24-48 hours, and 48-72 hours post-dose
Population: as for outcome 31
Measure: Mean (Standard Deviation); unit: Nanogram per hour (ng/h)
Arm/Group | Therapeutic Dose: ITF2357 100 mg | Supratherapeutic Dose: ITF2357 300 mg
Number analyzed (Participants) | 12 | 12
Nanogram per hour (ng/h)
  ITF2357 | 304920.74 (327302.13) | 1224735.12 (922878.78)
  ITF2374 | 155698.10 (166313.02) | 536094.03 (361645.28)
  ITF2375 | 51562.37 (46045.34) | 182276.01 (172602.20)
  ITF2440 | 1323571.78 (414580.11) | 3469056.76 (1554749.72)
  ITF2563 | 712846.46 (298304.19) | 1986177.40 (904296.76)
  ITF2955 glucuronide | 5170.46 (4743.78) | 25858.22 (23838.45)

33. Secondary Outcome: Urine PK: Time of Rmax (TRmax) for ITF2357 and Its Metabolites
Description: TRmax was calculated as the midpoint of the collection interval during which Rmax occurred for ITF2357 and Metabolites: ITF2374, ITF2375, ITF2440, ITF2563, ITF2955 glucuronide.
Time Frame: Pre-dose (within 2 hours before dosing), 0-8 hours, 8-24 hours, 24-48 hours, and 48-72 hours post-dose
Population: as for outcome 31
Measure: Median (Full Range); unit: hours
Arm/Group | Therapeutic Dose: ITF2357 100 mg | Supratherapeutic Dose: ITF2357 300 mg
Number analyzed (Participants) | 12 | 12
hours
  ITF2357 | 1.84 [0.34 to 3.77] | 1.49 [0.36 to 9.39]
  ITF2374 | 4.40 [0.34 to 11.01] | 1.49 [0.36 to 10.01]
  ITF2375 | 1.84 [0.34 to 10.01] | 1.49 [0.36 to 9.39]
  ITF2440 | 7.24 [0.34 to 11.01] | 6.65 [0.36 to 22.17]
  ITF2563 | 7.24 [0.34 to 11.01] | 6.65 [0.36 to 10.01]
  ITF2955 glucuronide | 1.84 [0.34 to 3.77] | 1.49 [0.36 to 3.79]

34. Secondary Outcome: Urine PK: Renal Clearance (Clr) for ITF2357 and Its Metabolites
Description: Clr was calculated as Ae0-t / AUC0-t (plasma) for ITF2357 and Metabolites: ITF2374, ITF2375, ITF2440, ITF2563, ITF2955 glucuronide.
Time Frame: Pre-dose (within 2 hours before dosing), 0-8 hours, 8-24 hours, 24-48 hours, and 48-72 hours post-dose
Population: The PK population was defined as all participants who completed at least 3 periods, including at least Treatments T, ST, and M for whom the PK profile was adequately characterized. Here, "Overall Number of Participants Analyzed" signifies participants evaluable for this outcome measure and "Number Analyzed" signifies participants evaluable at specific category.
Measure: Mean (Standard Deviation); unit: L/h
Arm/Group | Therapeutic Dose: ITF2357 100 mg | Supratherapeutic Dose: ITF2357 300 mg
Number analyzed (Participants) | 12 | 12
L/h
  ITF2357 | 2127.55 (402.63) | 1859.30 (360.82)
  ITF2374 | 3856.29 (979.36) | 3403.49 (1004.83)
  ITF2375 | 103.35 (27.94) | 96.02 (29.26)
  ITF2440 | 3629.92 (717.29) | 2994.15 (583.57)
  ITF2563 | 7879.16 (1464.33) | 7666.41 (1279.54)
  ITF2955 glucuronide: number analyzed (Participants) | 4 | 12
  ITF2955 glucuronide | 16623.97 (22459.53) | 4215.01 (1176.29)

35. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) and Serious TEAEs
Description: Adverse event (AE) was defined as any untoward medical occurrence in a subject or clinical investigation participant administered a pharmaceutical product and which did not necessarily have a causal relationship with the study drug. Serious adverse event (SAE) was an AE that resulted in any of the following outcomes: death; life threatening; persistent/significant disability/incapacity; required initial or prolonged inpatient hospitalization; congenital anomaly/birth defect or was otherwise considered medically important. TEAE were defined as an AEs following the start of treatment or AEs increasing in severity during treatment. TEAEs include both serious and non-serious TEAEs.
Time Frame: Baseline up to 44 days
Population: The Safety population was defined as all participants who received at least 1 dose of study drug (therapeutic and supratherapeutic doses of ITF2357, moxifloxacin, or placebo).
Measure: Count of Participants; unit: Participants
Arm/Group | Therapeutic Dose: ITF2357 100 mg | Supratherapeutic Dose: ITF2357 300 mg | Placebo | Moxifloxacin
Number analyzed (Participants) | 29 | 31 | 31 | 31
Participants
  Participants with TEAEs | 5 | 15 | 4 | 6
  Participants with Serious TEAEs | 0 | 0 | 0 | 0

36. Secondary Outcome: Number of Treatment-Related TEAEs
Description: Adverse event (AE) was defined as any untoward medical occurrence in a subject or clinical investigation participant administered a pharmaceutical product and which did not necessarily have a causal relationship with the study drug. Any AEs which occurred due to study drug treatment are reported as Treatment-related AEs. Number of treatment related TEAEs were reported.
Time Frame: Baseline up to 44 days
Population: as for outcome 35
Measure: Number; unit: number of events
Arm/Group | Therapeutic Dose: ITF2357 100 mg | Supratherapeutic Dose: ITF2357 300 mg | Placebo | Moxifloxacin
Number analyzed (Participants) | 29 | 31 | 31 | 31
number of events | 6 | 20 | 6 | 4

37. Secondary Outcome: Number of TEAEs Based on Severity
Description: All AEs were analyzed using National Cancer Institute-Common Terminology Criteria for Adverse Events (NCI-CTCAE) Version 5.0 and were graded as Grade 1: mild asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated, Grade 2: Moderate; minimal, local or noninvasive intervention indicated; limiting age-appropriate instrumental activities of daily living (ADL), Grade 3: Severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self care ADL, Grade 4: Life-threatening consequences; urgent intervention indicated, Grade 5: death related AE, where higher grade indicated more severe condition. Number of TEAEs based on severity were reported.
Time Frame: Baseline up to 44 days
Population: as for outcome 35
Measure: Number; unit: number of events
Arm/Group | Therapeutic Dose: ITF2357 100 mg | Supratherapeutic Dose: ITF2357 300 mg | Placebo | Moxifloxacin
Number analyzed (Participants) | 29 | 31 | 31 | 31
number of events
  Mild | 6 | 21 | 8 | 6
  Moderate | 0 | 4 | 0 | 0
  Severe | 0 | 0 | 0 | 0

38. Secondary Outcome: Number of Participants With Clinically Significant Changes in Vital Signs
Description: Vital signs, including semi supine blood pressure, pulse rate, respiratory rate, weight, and oral temperature were assessed. Clinical significance was decided by the investigator. Number of participants with clinically significant change from baseline in vital signs were reported.
Time Frame: Baseline up to 44 days
Population: as for outcome 35
Measure: Count of Participants; unit: Participants
Arm/Group | Therapeutic Dose: ITF2357 100 mg | Supratherapeutic Dose: ITF2357 300 mg | Placebo | Moxifloxacin
Number analyzed (Participants) | 29 | 31 | 31 | 31
Participants | 0 | 0 | 0 | 0

39. Secondary Outcome: Number of Participants With Clinically Significant Changes in Clinical Laboratory Parameters
Description: Clinical laboratory parameters included biochemistry, hematology, and urinalysis. Clinical significance was decided by the investigator. Number of participants with clinically significant change from baseline in clinical laboratory parameters were reported.
Time Frame: Baseline up to 44 days
Population: as for outcome 35
Measure: Count of Participants; unit: Participants
Arm/Group | Therapeutic Dose: ITF2357 100 mg | Supratherapeutic Dose: ITF2357 300 mg | Placebo | Moxifloxacin
Number analyzed (Participants) | 29 | 31 | 31 | 31
Participants | 0 | 2 | 0 | 0

40. Secondary Outcome: Number of Participants With Clinically Significant Changes in Electrocardiogram (ECG) Findings
Description: ECG parameters included rhythm, ventricular rate, PR interval, QRS duration, and QT interval. Clinical significance was decided by the investigator. Number of participants with clinically significant change from baseline in ECG were reported.
Time Frame: Baseline up to 44 days
Population: as for outcome 35
Measure: Count of Participants; unit: Participants
Arm/Group | Therapeutic Dose: ITF2357 100 mg | Supratherapeutic Dose: ITF2357 300 mg | Placebo | Moxifloxacin
Number analyzed (Participants) | 29 | 31 | 31 | 31
Participants | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Baseline up to 44 days
Description: The Safety population was defined as all participants who received at least 1 dose of study drug (therapeutic and supratherapeutic doses of ITF2357, moxifloxacin, or placebo).
Arm/Group | Therapeutic Dose: ITF2357 100 mg | Supratherapeutic Dose: ITF2357 300 mg | Placebo | Moxifloxacin
All-Cause Mortality (participants affected / at risk) | 0/29 | 0/31 | 0/31 | 0/31
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/31 | 0/31 | 0/31
Other Adverse Events (participants affected / at risk) | 5/29 | 15/31 | 6/31 | 4/31
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Therapeutic Dose: ITF2357 100 mg (N=29) | Supratherapeutic Dose: ITF2357 300 mg (N=31) | Placebo (N=31) | Moxifloxacin (N=31)
Nausea (Gastrointestinal disorders) | 0 (0) | 5 (5) | 0 (0) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 1 (1) | 2 (2) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Eructation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Faeces soft (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 4 (4) | 1 (1) | 0 (0)
Disturbance in attention (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
White blood cells urine positive (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Blood triglycerides increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Heart rate irregular (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sensation of foreign body (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vessel puncture site haematoma (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Folliculitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-09-29): https://cdn.clinicaltrials.gov/large-docs/63/NCT04821063/Prot_000.pdf
  • Statistical Analysis Plan (2021-06-11): https://cdn.clinicaltrials.gov/large-docs/63/NCT04821063/SAP_001.pdf